CLINICAL TRIAL: NCT03507881
Title: Prospective Study on Clinical and Radiological Results With Ennovate® Pedicle Screw Fixation in Isthmic Spondylolisthesis Patients
Brief Title: Prospective Study on Ennovate® Pedicle Screw Fixation in Isthmic Spondylolisthesis Patients
Acronym: ENNOVIST
Status: Terminated | Type: Observational
Why Stopped: Recruitment too slow
Sponsor: Aesculap AG (Industry)
Collaborators: Raylytic GmbH (Industry); ZKS Münster (Unknown)
Responsible Party: Sponsor
Other Study IDs: AAG-O-H-1619
Record Dates: First submitted 2018-04-16; First posted 2018-04-25 (Actual); Last update posted 2019-09-18 (Actual); Status verified 2019-09

CONDITIONS: Spine Fusion; Isthmic Spondylolisthesis
Keywords: isthmic spondylolisthesis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ennovate: Implantation of an Ennovate® internal fixation
  Interventions: Device: fusion

INTERVENTIONS:
Device: fusion — Internal fixation

SUMMARY:
The present study is planned to demonstrate the efficacy and safety of a new pedicle screw system for the specific indication of isthmic spondylolisthesis, as this condition concerns relatively young patients requiring good fixation of the performed reposition to come to satisfactory clinical results.

DETAILED DESCRIPTION:
Adult Isthmic spondylolisthesis, which is associated with "spondylolysis," is defined as an osseous discontinuity of the vertebral arch at the isthmus (the pars interarticularis), which usually occurs in the fifth lumbar vertebra. The prevalence of isthmic spondylosis is proposed to be about 6% to 26% in different studies. The European Spine Tango registry found 15%. It is proposed to affect more men than women. Conservative treatments including braces, physical therapy, and medication are shown to be effective for some patients; however, surgical treatments are mainly the final effective treatment. There are several different options for surgery among which posterolateral fusion (PLF) is considered as the method of choice. It is shown that PLF is more effective than conservative treatments such as exercise. The fusion helps to fix the motion of the affected segment and therefore, might lead to pain reduction. Decompression, supplemental instrumentation, and supplemental anterior column support are also considered for treatment. These treatment strategies can be used separately or in any combination; however, studies trying to compare separate treatments with a combination of them have led to inconsistent results.

Supplementary pedicle screws might be added to fusion methods for fixation and it is proposed that they have the ability to correct the deformity, reduce the listhesis, and increase the fusion rates, although a majority of the studies comparing instrumented PLF and noninstrumented PLF could not show the superiority of instrumented approaches. The literature has been reviewed in 2000 already, and the method has already been proved to be "practical, safe, and effective" for various spinal indications. Other authors found a better result for isthmic spondylolisthesis patients with posterior lumbar interbody Fusion (PLIF), vs. PLF, especially for high grade isthmic spondylolisthesis.

The present study is planned to demonstrate the efficacy and safety of a new pedicle screw system for the specific indication of isthmic spondylolisthesis, as this condition concerns relatively young patients requiring good fixation also in the long-term.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic single-level IS (L4-S1), (VAS > 30mm, treated conservatively for a minimum of 6 months)
* Isthmic Spondylolisthesis Meyerding grade I and II
* Signed Informed Consent of the patient regarding the participation in this study

Exclusion Criteria:

* Multilevel IS
* Severe degenerative changes of cranial adjacent level (disc height of <50% of the next healthy segment,
* Previous lumbar spine surgery except microdiscectomy or micro- decompression of the index level
* Patients psychically or mentally not able to give or refuse consent
* Patients psychically or mentally not able to answer the questions regarding their health status and quality of life
* Pregnancy (current or planned)
* BMI >35
* Systemic or local infection
* Chemotherapy or radiation ongoing
* Desire of early retirement (running pension request)
* All contraindications as listed in the instructions for use

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult patients
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2018-07-31 (Actual); Primary Completion 2019-01-18 (Actual); Study Completion 2019-01-18 (Actual)

PRIMARY OUTCOMES:
Leg pain | 1 year
  Leg Pain measured by Visual analogue scale (VAS) after 1 year follow-up: measured by Visual Analogue Scale: The visual analogue scale or visual analog scale (VAS) is a psychometric response scale which can be used in questionnaires. It is a measurement instrument for subjective characteristics or attitudes that cannot be directly measured. When responding to a VAS item, respondents specify their level of agreement to a statement by indicating a position along a continuous line between two end-points.

SECONDARY OUTCOMES:
Leg Pain | Preoperative, 3 months, 6 months
  Leg Pain measured by Visual analogue scale (VAS) at all timepoints except 1 year; measured by Visual Analogue Scale: The visual analogue scale or visual analog scale (VAS) is a psychometric response scale which can be used in questionnaires. It is a measurement instrument for subjective characteristics or attitudes that cannot be directly measured. When responding to a VAS item, respondents specify their level of agreement to a statement by indicating a position along a continuous line between two end-points.
Back Pain | Preoperative, 3 months, 6 months, 1 year
  Back Pain measured by Visual analogue scale (VAS) at all timepoints; measured by Visual Analogue Scale: The visual analogue scale or visual analog scale (VAS) is a psychometric response scale which can be used in questionnaires. It is a measurement instrument for subjective characteristics or attitudes that cannot be directly measured. When responding to a VAS item, respondents specify their level of agreement to a statement by indicating a position along a continuous line between two end-points.
Functional Disability | Preoperative, 3 months, 6 months, 1 year
  Measured by Oswestry Disability Index (ODI) at all timepoints; The ODI is an index derived from the Oswestry Low Back Pain Questionnaire to quantify disability for low back pain. The self-completed questionnaire contains ten Topics: intensity of pain, lifting, ability to care for oneself, ability to walk, ability to sit, sexual function, ability to stand, social life, sleep quality, and ability to travel. Each topic category is followed by 6 statements describing different potential scenarios in the patient's life relating to the topic. Each question is scored on a scale of 0-5 with the first statement being zero and indicating the least amount of disability and the last statement is scored 5 indicating most severe disability. The scores for all questions answered are summed, then multiplied by two to obtain the index (range 0 to 100). Zero is equated with no disability and 100 is the maximum disability possible.
Patient satisfaction | 3 months, 6 months, 1 year
  Patient Satisfaction with Operation Result (very high / high / medium / low / very low)
Quality of Life | preoperative, 3 months, 6 months, 1 year
  Quality of Life measured by EQ-5D-5L Questionnaire: The 5-level EQ-5D version (EQ-5D-5L) was introduced by the EuroQol Group in 2009 to improve the instrument's sensitivity and to reduce ceiling effects, as compared to the EQ-5D-3L. The EQ-5D-5L essentially consists of 2 pages: the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS). The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety / depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
Clinical Complications | intraoperative, 3 months, 6 months, 1 year
  Adverse Events (AE) and Serious Adverse Events (SAE) forms filled at all timepoints intraop and postop
Fusion status | 3 months, 6 months, 1 year
  Fusion assessment (acc. to Bridwell)
Radiographically assessed complications | 3 months, 6 months, 1 year
  Construct stability, loosening, implant breakage, other adverse events (Osteolysis, screw misplacement, device migration)
Loss of Reduction of the Reposition [degree] | 3 months, 6 months, 1 year
  Results regarding the maintenance of the reposition of the isthmic spondylolisthesis throughout the follow-up; loss of reduction during follow-up measured in [degree]
Range of Motion | 3 months, 6 months, 1 year
  Range of motion (angular and translational; degrees/mm)

CONTACTS AND LOCATIONS:
Locations (3):
- Germany (3):
  - Klinikum der J. W. Goethe-Universität, Klinik für Allgemein- und Visceralchirurgie, Frankfurt am Main
  - Katholisches Klinikum Koblenz, Koblenz
  - Sana Klinikum Offenbach GmbH, Offenbach

REFERENCES:
- [Background] Gaines RW Jr. The use of pedicle-screw internal fixation for the operative treatment of spinal disorders. J Bone Joint Surg Am. 2000 Oct;82(10):1458-76. doi: 10.2106/00004623-200010000-00013. PMID 11057475
- [Background] Dehoux E, Fourati E, Madi K, Reddy B, Segal P. Posterolateral versus interbody fusion in isthmic spondylolisthesis: functional results in 52 cases with a minimum follow-up of 6 years. Acta Orthop Belg. 2004 Dec;70(6):578-82. PMID 15669459
- [Background] Etemadifar MR, Hadi A, Masouleh MF. Posterolateral instrumented fusion with and without transforaminal lumbar interbody fusion for the treatment of adult isthmic spondylolisthesis: A randomized clinical trial with 2-year follow-up. J Craniovertebr Junction Spine. 2016 Jan-Mar;7(1):43-9. doi: 10.4103/0974-8237.176623. PMID 27041885
- [Background] Taillard WF. Etiology of spondylolisthesis. Clin Orthop Relat Res. 1976 Jun;(117):30-9. PMID 1277680
- [Background] Kalichman L, Kim DH, Li L, Guermazi A, Berkin V, Hunter DJ. Spondylolysis and spondylolisthesis: prevalence and association with low back pain in the adult community-based population. Spine (Phila Pa 1976). 2009 Jan 15;34(2):199-205. doi: 10.1097/BRS.0b013e31818edcfd. PMID 19139672
- [Background] McTimoney CA, Micheli LJ. Current evaluation and management of spondylolysis and spondylolisthesis. Curr Sports Med Rep. 2003 Feb;2(1):41-6. doi: 10.1249/00149619-200302000-00008. PMID 12831675
- [Background] STEWART TD. [The age incidence of neural-arch defects in Alaskan natives, considered from the standpoint of etiology]. J Bone Joint Surg Am. 1953 Oct;35-A(4):937-50. No abstract available. Undetermined Language. PMID 13108895
- [Background] Osterman K, Schlenzka D, Poussa M, Seitsalo S, Virta L. Isthmic spondylolisthesis in symptomatic and asymptomatic subjects, epidemiology, and natural history with special reference to disk abnormality and mode of treatment. Clin Orthop Relat Res. 1993 Dec;(297):65-70. PMID 8242953
- [Background] Jacobs WC, Vreeling A, De Kleuver M. Fusion for low-grade adult isthmic spondylolisthesis: a systematic review of the literature. Eur Spine J. 2006 Apr;15(4):391-402. doi: 10.1007/s00586-005-1021-4. Epub 2005 Oct 11. PMID 16217665
- [Background] GILL GG, MANNING JG, WHITE HL. Surgical treatment of spondylolisthesis without spine fusion; excision of the loose lamina with decompression of the nerve roots. J Bone Joint Surg Am. 1955 Jun;37-A(3):493-520. No abstract available. PMID 14381447
- [Background] France JC, Yaszemski MJ, Lauerman WC, Cain JE, Glover JM, Lawson KJ, Coe JD, Topper SM. A randomized prospective study of posterolateral lumbar fusion. Outcomes with and without pedicle screw instrumentation. Spine (Phila Pa 1976). 1999 Mar 15;24(6):553-60. doi: 10.1097/00007632-199903150-00010. PMID 10101819
- [Background] Moller H, Hedlund R. Instrumented and noninstrumented posterolateral fusion in adult spondylolisthesis--a prospective randomized study: part 2. Spine (Phila Pa 1976). 2000 Jul 1;25(13):1716-21. doi: 10.1097/00007632-200007010-00017. PMID 10870149
- [Background] Thomsen K, Christensen FB, Eiskjaer SP, Hansen ES, Fruensgaard S, Bunger CE. 1997 Volvo Award winner in clinical studies. The effect of pedicle screw instrumentation on functional outcome and fusion rates in posterolateral lumbar spinal fusion: a prospective, randomized clinical study. Spine (Phila Pa 1976). 1997 Dec 15;22(24):2813-22. doi: 10.1097/00007632-199712150-00004. PMID 9431617
- [Background] McGuire RA, Amundson GM. The use of primary internal fixation in spondylolisthesis. Spine (Phila Pa 1976). 1993 Sep 15;18(12):1662-72. doi: 10.1097/00007632-199309000-00015. PMID 8235847